CLINICAL TRIAL: NCT04579276
Title: Different Approaches to Thoracic Paravertebral Block: a Monocentric Randomized Study Comparing Ultrasounded-guided Method to Intrathoracic Visual Method
Brief Title: Different Approaches to Thoracic Paravertebral Block
Acronym: VAP BLOCK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020-11; 2020-A00483-36 (Other: IDRCB)
Record Dates: First submitted 2020-09-04; First posted 2020-10-08 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Thoracotomy
MeSH Terms: interventions — Tea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "surgical" method (Experimental)
  Interventions: Procedure: Thoracic paravertebral block
- "anesthetic" method (Active Comparator)
  Interventions: Procedure: thoracic epidural analgesia

INTERVENTIONS:
Procedure: Thoracic paravertebral block — Intrathoracic method undergone through video assisted surgery (VATS
  Arms: "surgical" method
Procedure: thoracic epidural analgesia — locoregional analgesia under ultrasound control
  Arms: "anesthetic" method

SUMMARY:
Thoracic paravertebral block (TPB) in thoracic surgery is practiced since the development of minimally invasive surgery. Historically, thoracic epidural analgesia is done in open thoracic surgery. Thoracotomy with rib spacing causes strong post-operative pain that is well controlled with epidural analgesia and allows less use of morphine. However, this method causes frequent side effects. Minimally invasive surgery, when it is possible and recommended, has the main benefit of not spacing the ribs and therefore preventing nerve stretching, rib fractures and less post-operative pain. This less aggressive method has other benefits: less inflammation, better recuperation especially for vulnerable patients (the elderly; limited pulmonary functions), less time of thoracic drainage, less in hospital stay and better quality of life (1). Less invasive surgery has brought us to use less invasive analgesic methods. Thoracic paravertebral block is a good alternative to thoracic epidural analgesia but is unfortunately not done everywhere due to the lack and need of professional training. The objective of our study is to compare two methods of TPB: ultrasound guided method undergone by the anesthesiologist, and intrathoracic method undergone through video assisted surgery (VATS) or robotic assisted surgery (RATS).

DETAILED DESCRIPTION:
A randomized prospective mono-centric non-inferiority controlled and simple blinded study comparing the "surgical" method (experimental group) to the "anesthetic" method (control group) for patients operated in thoracic minimally invasive surgery (VATS or RATS).

Recruitment: Patients undergoing therapeutic or diagnostic surgery in the thoracic ward of the university hospital of Marseille.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age.
* VATS or RATS with lung resection including wedges, segmentectomies or lobectomies.
* Signed consent.
* Scheduled surgeries.

Exclusion Criteria:

* Patient refusing to sign the consent form.
* Minors.
* Patients under any guardianship.
* All surgeries with pleura intervention: talc, pleurectomy, wall resection.
* Non trained anesthesiologist to ultrasound TPB.
* Presence of pain or daily use of painkillers prior to surgery.
* Medical history of homolateral thoracic surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
total morphine consumption | 48 HOURS

SECONDARY OUTCOMES:
Time occupancy of the operating room | 1 MONTH
visual analog scale of pain (VAS) | 12 HOURS
visual analog scale of pain (VAS) | 48HOURS
visual analog scale of pain (VAS) | 30 DAYS

CONTACTS AND LOCATIONS:
Overall Officials: Emilie GARRIDO- PRADALIE, Study Director — Assistance Publique Hopitaux De Marseille; JOSEPHINE CHENESSEAU, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- assistance publique hôpitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Chenesseau J, Fourdrain A, Pastene B, Charvet A, Rivory A, Baumstarck K, Bouabdallah I, Trousse D, Boulate D, Brioude G, Gust L, Vasse M, Braggio C, Mora P, Labarriere A, Zieleskiewicz L, Leone M, Thomas PA, D'Journo XB. Effectiveness of Surgeon-Performed Paravertebral Block Analgesia for Minimally Invasive Thoracic Surgery: A Randomized Clinical Trial. JAMA Surg. 2023 Dec 1;158(12):1255-1263. doi: 10.1001/jamasurg.2023.5228. PMID 37878299